CLINICAL TRIAL: NCT06370065
Title: Efficacy and Safety of Serplulimab Combined With Bevacizumab Biosimilar and HAIC in Advanced Hepatocellular Carcinoma (HCC) Patients
Brief Title: Serplulimab Combined With Bevacizumab Biosimilar and HAIC in Advanced Hepatocellular Carcinoma (HCC) Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT70-TJ
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC+Serplulimab（HLX10）+ Bevacizumab Biosimilar（HLX04） (Experimental): Procedure: HAIC (Hepatic arterial infusion chemotherapy) Drug: HLX10 (PD-1 antibody) Drug: HLX04 (VEGF antibody) HAIC: FOLFOX, q3w, up to 8 times; HLX10: 4.5mg/kg, iv, q3w, ; HLX04: 10mg/kg, iv, q3w.
  Interventions: Drug: HAIC+Serplulimab（HLX10）+ Bevacizumab Biosimilar（HLX04）

INTERVENTIONS:
Drug: HAIC+Serplulimab（HLX10）+ Bevacizumab Biosimilar（HLX04） — PD-1 inhibitor

SUMMARY:
Evaluation of the efficacy and safety of Serplulimab combined with bevacizumab biosimilar and HAIC in Advanced Hepatocellular Carcinoma (HCC) patients

ELIGIBILITY:
Inclusion Criteria:

1. Willing to attend the study and having given the ICF
2. Age ≥18
3. Have a HCC diagnosis confirmed by radiology, histology, or cytology HCC is diagnosed at Barcelona Clinic Liver Cancer (BCLC) Stage C
4. Have not accepted any of systemic therapy for HCC such as systemic chemotherapy, molecular targeted drugs, immunotherapy.
5. At least 1 measurable intrahepatic lesion suitable for repeat assessments according to RECISTv1.1 criteria and it has not undergone surgery, radiology and/or other regional therapy (including but not limited to radiofrequency ablation, percutaneous ethanol injection, freezing therapy, high intensity focused ultrasound, transcatheter arterial chemoembolization, transcatheter arterial embolization). But if it progressed after the regional therapy, it could be selected as a target lesion. The local regional therapy must be done 4 weeks before randomization and the related AEs must recover to ≤ CTCAE grade 1.
6. Child-Pugh score ≤7
7. Eastern Cooperative Oncology Group (ECOG) 0 or 1
8. Expected life time is over 12 weeks.
9. HBV-DNA < 2000 IU/mL
10. Organs function:

Platelet count ≥75×109/L Absolute neutrophil count (ANC) ≥1.5×109 /L White blood cell count ≥3.0×109 /L Haemoglobin ≥9.0 g/dL Serum total bilirubin ≤1.5×ULN ALT ≤5×ULN, and AST ≤5×ULN（ALT ≤3×ULN, and AST ≤3×ULN, if HCV-RNA is detectable） Albumin ≥28 g/L INR ≤1.5×ULN PT ≤1.5×ULN APTT ≤1.5×ULN Creatinine clearance (CL) >50 mL/min or serum creatinine ≤1.5×ULN Urine protein ≤1+ or ≤1.0g/24h 12. Patient is not fertile or willing and able to obey effective contraception

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma and HCC
2. History of hepatic encephalopathy
3. History of GI bleeding within 6 months, or investigator defined with high risk of haemorrhage for esophageal varices
4. With distant metastasis (hilar lymph nodes metastasis is allowed)
5. Co-infection of HBV and HCV
6. History of other malignancy within 5 years except for healed local tumor.
7. History of or plan to accept allogenic organ transplantation
8. Ascites requiring invasive intervention (e.g. paracentesis) to maintain symptomatic control (every month or more often)
9. History of myocardial infarction or unstable angina or uncontrolled arrythmia or stroke or cerebral hemorrhage within 6 months prior to randomization. QTcF value ≥450ms（male）or ≥470ms（female） detected by 12-lead electrocardiogram.
10. New York Heart Association Grade ≥2 congestive heart failure or LVEF <50%
11. Uncontrolled hypertension
12. History of hypertensive crisis or hypertensive encephalopathy
13. Active infection including but not limited to tuberculosis and HIV
14. With interstitial lung disease, lung fibrosis, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia and serious impairment in lung function
15. Active autoimmune disorders except patients with substitutional treatment with thyroid hormone and type I diabetes under treatment with insulin.
16. Receipt of live attenuated vaccine within 28 days prior to randomization
17. Current or prior use of steroids (>10mg/d prednisone) or immunosuppressive medication within 14 days before randomization
18. Significant traumatic injury or major surgical procedure within 28 days prior to randomization
19. Receipt of checkpoint inhibitors or T cell costimulatory drugs
20. Receipt of bevacizumab or its analogues
21. Involved in another clinical trial less than 14 days before randomization
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
23. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control
24. Active bleeding, with history of ≥grade 3 bleeding within 6 months, or ≥grade 2 bleeding within 3 months
25. Use of anti-thrombotics within 5 days prior to randomization
26. In need of NSAIDs for long-term treatment.

26.With one of the following diseases within 6 months before randomization:(1) Digestive fistula, perforation and abscess (2) Gastrointestinal obstruction (3) Abdominal infection or inflammation (4) Major vascular disease 28. With severe and green wound, active ulcer or untreated fracture 29. History of drug abuse 30. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to screen for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 1year
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
PFS | up to 1 year
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
OS | up to 2 years
  Defined as the time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol